CLINICAL TRIAL: NCT01170052
Title: Phase I/II Study With Bendamustine and Temsirolimus in Patients With Relapsed or Refractory Mantle Cell Non-hodgkin's Lymphoma (NHL) Not Eligible for High Dose Chemotherapy and Autologous/Allogeneic Stem Cell Transplantation
Brief Title: Bendamustine and Temsirolimus in Patients With Relapsed or Refractory Mantle Cell Non-Hodgkin's Lymphoma (NHL)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Mundipharma K.K. (Industry)
Responsible Party: Principal Investigator: Christian Scholz, PD Dept. of Hematology, Charité Berlin, Germany, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-No.: 2009-014844-13
Record Dates: First submitted 2010-07-14; First posted 2010-07-27 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2010-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: Relapsed Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma; Non-Hodgkins Lymphoma; Temsirolimus; Bendamustine; Phase 1/2
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — temsirolimus; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus 75mg i.v. day 1, 8, 15, 21 for a 28 day cycle with a maximum of 6 Cycles.
  Other Names: Torisel®
Drug: Bendamustine — Bendamustin 90mg/m2 i.v. day 2 and 3 for a 28 day cycle with a maximum of 6 Cycles.
Drug: Temsirolimus — Consolidation Therapy for Patients reached CR or PR with Temsirolimus 75mg weekly until progression.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and activity of the combination of bendamustine and rituximab in patients with relapsed/refractory mantle cell lymphoma who are not eligible for high dose chemotherapy and autologous/allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Mantle Cell Lymphoma according to REAL/WHO classification
* First or second relapse or alternatively progression during therapy. Previous use of Bendamustine is permitted, if the patient has reached at least partial remission and progression occured more than 6 months after therapy. Previous high dose chemotherapy with auto-SCT is permitted, if the patient has reached at least partial remission and progression occured more than 12 months after therapy.
* Patients must not be eligible for high dose chemotherapy with auto-SCT or allo-SCT.
* Adequate bone marrow function (hemoglobin > 9g/dl, platelet count >100/nL, absolute neutrophil count >1,5 /nL)
* WHO/ECOG Performance Status 0-2
* Measurable disease (two perpendicular diameters by either physical or radiological examination)
* Life expectancy ≥ 3 weeks
* Written informed consent

Exclusion Criteria:

* Prior treatment with any m-TOR Inhibitor
* Unstable or severe uncontrolled medical condition (e.g. severe congestive heart failure, myocardial infarction within the past 6 months, severe, uncontrolled arterial hypertension, renal insufficiency requiring hemodialysis, severe pulmonary disease, severe diabetes)
* Abnormal liver function: transaminases or total bilirubin > 2 x upper limit of normal (ULN)
* Abnormal renal function: serum creatinine > 2 x upper limit of normal
* Previous malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix.
* Concurrent treatment with strong inhibitors of CYP3A4 and/or inducers of CYP3A4
* Pregnant or breastfeeding women (negative pregnancy test not older than 7 days is required for women of fertile age). Men and women of child-bearing potential must agree to use adequate contraception (i.e. failure rate < 1% p.a. )
* Major surgery within 4 weeks before study entry; minor procedures (e.g. Implantation i.v. port catheter, Lymphnode biopsy) within 1 week before study entry
* Previous therapy with any investigational agents within 28 days before study entry
* Concomitant immunotherapy (e.g. Rituximab) or Chemotherapy other than Bendamustine. Use of systemic steroids should be documented and the Principal Investigator be informed.
* Central nervous system (CNS) lymphomatous involvement
* HIV positivity
* Current or chronic hepatitis B or hepatitis C infection
* Severe psychiatric illness or Individuals that are placed in an institution due to a magisterial or judiciary command.
* Inability to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose-finding | 6 months
  Is the combination of temsirolimus alongside with bendamustine at the suggested dose feasible or are dose reductions necessary. Number of dose reductions or delays of therapy due to hematologic toxicities (CTCAE) or other adverse events according to protocoll.
Phase II: Response Rate (Overall response rate, complete and partial response) | 6 months
  What is the response rate of a therapy with temsirolimus and bendamustine.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  This is defined as the period of time between the admission into the clinical trial and the progression of the lymphoma or death of any kind.
Safety and Tolerability of Temsirolimus and Bendamustine Combination Therapy | 2 years
  Detection of overall toxicity, serious adverse events (SAE), suspected unexpected serious adverse reactions (SUSAR) during treatment with temsirolimus and bendamustine.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Scholz, PD Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (3):
- Germany (3):
  - Dept. of Hematology and Oncology, Charité, Campus Charité Mitte, Berlin, State of Berlin
  - Dept. of Hematology and Oncology, Charité, Campus Benjamin Franklin, Berlin, State of Berlin
  - Dept. of Hematology and Oncology, Charité, Campus Virchow Klinikum Charité, Berlin, State of Berlin